CLINICAL TRIAL: NCT02090179
Title: Evaluation of Blood Brain Barrier Integrity and Relationship to Structural Brain Abnormalities in MPS IIIB Patients Using Cerebrospinal Fluid/Serum Albumin Index (CSF-AI) and Multimodal Magnetic Resonance Imaging
Brief Title: Evaluation of Blood Brain Barrier Integrity and Structural Abnormalities in MPS IIIB Patients Using Multimodal Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NGLU-CL01; 2013-001938-18 (EudraCT Number)
Record Dates: First submitted 2014-03-12; First posted 2014-03-18 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: MPS IIIB (Sanfilippo B Syndrome)
Keywords: MPS IIIB; Mucopolysaccharidosis; Mucopolysaccharidosis type IIIB; Sanfilippo Syndrome; Metabolism, Inborn Errors; Metabolic Diseases; Genetic Diseases, Inborn
MeSH Terms: conditions — Mucopolysaccharidosis III; Mucopolysaccharidoses; Metabolism, Inborn Errors; Metabolic Diseases; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MPS IIIB: Those with a definitive diagnosis of MPS IIIB (Sanfilippo B Syndrome).

SUMMARY:
The purpose of the study is to characterize structural abnormalities in the brain and the integrity of the blood brain barrier in patients with mucopolysaccharidosis type IIIB (MPS IIIB).

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or subject's parent or legal guardian provides informed consent
* Subject is ≥5 years of age.
* Subject has a definitive diagnosis of MPS IIIB, as determined by either a documented deficiency in alpha-N-acetylglucosaminidase (NAGLU) enzyme activity or documented functionally-relevant mutations in both alleles of the NAGLU gene.

Exclusion Criteria:

* The subject has any internal or non-removable external metal items that may present a safety risk (for MRI), or any other medical condition or circumstance in which an MRI is contraindicated.
* The subject has a known or suspected hypersensitivity to anaesthesia, a bleeding disorder, or any other medical condition or circumstance in which a lumbar puncture (for collection of CSF) is contraindicated.
* Previous allergic reaction to gadolinium-based MRI contrast media.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to six subjects with MPS IIIB. An attempt will be made to enroll equal numbers (three) of MPS IIIB subjects with a classic (severe) disease presentation, and MPS IIIB subjects with an attenuated phenotype.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Blood Brain Barrier integrity in MPS IIIB subjects | Day 0
  Blood Brain Barrier integrity in MPS IIIB subjects by estimating the CSF-AI.
Blood Brain Barrier transfer coefficient | Day 0
  The Blood Brain Barrier transfer coefficient will be measured by DCE-MRI in MPS IIIB subjects.

SECONDARY OUTCOMES:
Structural brain abnormalities in MPS IIIB | Day 0
  Structural brain abnormalities in MPS IIIB using imaging and biomarkers related to underlying disease biology of MPS IIIB subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Birmingham, United Kingdom